CLINICAL TRIAL: NCT02268838
Title: A Phase 1 Single/ Multiple-Dose Study of E6007 in Healthy Japanese Male Subjects
Brief Title: Single/ Multiple-Dose Study of E6007 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6007-J081-002
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
Keywords: E6007; Healthy Japanese male subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 50 mg E6007 fasted condition (Experimental): E6007 50mg or E6007 matching placebo x 1, orally once daily in the morning under fasted condition. Drug administration on 1 day for single dose period (Day 1) and 7 days (Day 5 to 11) for repeated dose period.
  Interventions: Drug: E6007; Drug: E6007 matching placebo
- 100 mg E6007 fasted condition (Experimental): E6007 50mg or E6007 matching placebo x 2, orally once daily in the morning under fasted condition. Drug administration on 1 day for single dose period (Day 1) and 7 days (Day 5 to 11) for repeated dose period.
  Interventions: Drug: E6007; Drug: E6007 matching placebo
- 200 mg E6007 fasted condition (Experimental): E6007 50mg or E6007 matching placebo x 4, orally once daily in the morning under fasted condition. Drug administration on 1 day for single dose period (Day 1) and 7 days (Day 5 to 11) for repeated dose period.
  Interventions: Drug: E6007; Drug: E6007 matching placebo
- 400 mg E6007 fasted condition (Experimental): E6007 50mg or E6007 matching placebo x 8, orally once daily in the morning under fasted condition. Drug administration on 1 day for single dose period (Day 1) and 7 days (Day 5 to 11) for repeated dose period.
  Interventions: Drug: E6007; Drug: E6007 matching placebo
- 200 mg E6007 fed condition (Experimental): E6007 50mg or E6007 matching placebo x 4, orally once daily in the morning under fed condition. Drug administration on 1 day (Day 1).
  Interventions: Drug: E6007; Drug: E6007 matching placebo

INTERVENTIONS:
Drug: E6007
Drug: E6007 matching placebo

SUMMARY:
This is a single-center, placebo-controlled, randomized, ascending dose, double-blind study. This study will be evaluating ascending doses of 50, 100, 200, and 400 mg of E6007. This study consists of 5 steps, 1 to 5. In steps 1 to 4 (at ascending doses of 50, 100, 200, and 400 mg), subjects will be randomly assigned in a 6:2 ratio (E6007: placebo) to receive single dose of the study drug under fasted condition. Following 3 days of washout period, subject will receive the study drug once daily for 7 days starting on the fifth day from the single dose administration.

For step 3 (200 mg), subjects will subsequently have at least 17 days of washout period before being escalated to step 5 (200 mg) to receive single dose of E6007 under fed condition, to evaluate food effect of the study drug.

ELIGIBILITY:
Inclusion criteria

Subjects must meet all of the following criteria to be included in this study:

1. Healthy Japanese male subjects aged 20 to 44 years at the time of informed consent.
2. Has voluntarily consented, in writing, to participate in this study.
3. Has been thoroughly briefed on the conditions for participation in the study, and is willing and able to comply with the conditions.

Exclusion criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Has a clinically significant medical condition requiring treatment within 8 weeks before the initial study drug administration, or a history of clinically significant infection requiring treatment within 4 weeks before the initial drug administration.
2. History of surgical treatment such as resection of the liver, kidney, or Gastrointestinal tract, that may affect the Pharmacokinetic profiles of study drugs.
3. Ineligible for study participation in the opinion of the investigator or sub-investigator.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of E6007 as a measure of Adverse events | Screening and up to 17 days after last administration of drug
Plasma E6007 concentration over time period - Cmax (maximum concentration) | Up to 15 days
Plasma E6007 concentration over time period - tmax (Time to achieve maximum concentration (Cmax)) | Up to 15 days
Plasma E6007 concentration over time period - AUC (0-t) (Area Under the Curve (AUC) from Time Zero to Last Quantifiable Concentration) | Up to 15 days
Plasma E6007 concentration over time period - AUC (0-inf) (AUC extrapolated to infinity) | Up to 15 days
Plasma E6007 concentration over time period - t1/2 (Terminal phase half-life) | Up to 15 days
Plasma E6007 concentration over time period - CL/F (Apparent clearance) | Up to 15 days
Plasma E6007 concentration over time period - Vz/F (Apparent volume of distribution) | Up to 15 days
Plasma E6007 concentration over time period - Css,max (maximum steady state concentration) | Up to 15 days
Plasma E6007 concentration over time period - AUC (0-tau) (AUC from time zero to time tau over a dosing interval at steady state) | Up to 15 days

SECONDARY OUTCOMES:
Dose proportionality under fasted conditions with Cmax, AUC (0-t), AUC(0-inf), Cssmax and AUC(0-t) | Up to 15 days
Geometric mean proportion (fed:fasted) of Cmax, AUC(0-t) and AUC(0-inf) for 200mg E6007 dose | Up to 5 days
Evaluate relationship between E6007 plasma concentrations and electrocardiogram (ECG) parameter (QTcF) | Up to 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sumida-ku, Tokyo, Japan